CLINICAL TRIAL: NCT01989091
Title: Multi-Center, Prospective, Randomized, Open-Label, Sponsor-Blinded, Active-Control (Heparin) Clinical Investigation to Evaluate the Safety and Effectiveness of B-Lock™ as an Antimicrobial Catheter Lock Solution in Dialysis Patients With a Central Venous Catheter
Brief Title: Efficacy Study to Evaluate B-Lock™ as an Antimicrobial Lock Solution in Dialysis Patients With a CVC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Did not meet predetermined primary endpoint
Sponsor: Great Lakes Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GL-CL-0001
Record Dates: First submitted 2013-10-30; First posted 2013-11-20 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Dialysis Catheter Infections
Keywords: kidney dialysis; hemodialysis; locking solution; antimicrobial; thrombolytic
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B-Lock (IMD) (Experimental): Investigational Medical Device (IMD)
  Interventions: Device: B-Lock
- Heparin 5,000 U/mL (ACH) (Active Comparator): Active Comparator Heparin (ACH)
  Interventions: Drug: Heparin 5,000 U/mL

INTERVENTIONS:
Device: B-Lock — Antimicrobial Catheter Lock Solution
  Other Names: IMD
  Arms: B-Lock (IMD)
Drug: Heparin 5,000 U/mL — Standard of Care Catheter Lock Solution
  Other Names: ACH
  Arms: Heparin 5,000 U/mL (ACH)

SUMMARY:
Hypothesis: B-Lock is a safe and effective catheter lock solution that will maintain catheter patency and reduce Central Line Associated Blood Stream Infections (CLABSI) in dialysis patients using a central venous catheter (CVC) for vascular access.

The study is a prospective, randomized, site unblinded/sponsor blinded, clinical study of a minimum of 300 dialysis patients using a central venous catheter (CVC) for vascular access. Patients will be randomized 1:1 to receive either the investigational medical device (B-Lock or IMD) or active control heparin (5000 U/mL) (ACH) and observed for a minimum of 45 days or a maximum of 273 (expected average 160 days). IMD or ACH will be instilled into the catheter lumens (dual lumen catheters) at the end of each dialysis session and removed prior to the initiation of the next dialysis session.

The primary objectives of this study are:

* To demonstrate the safety of B-Lock in dialysis patients
* To demonstrate the non-inferiority or, if proven to be non-inferior, superiority of B-Lock relative to ACH with respect to maintaining catheter patency as defined by the use of recombinant tissue plasminogen activator for maintaining adequate blood flow through the dialysis catheter
* To demonstrate the superiority of B-Lock relative to ACH with respect to the incidence of CLABSI

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 18 to 80 years, inclusive. Patients, age 81 to 85 years, inclusive, may be included on a case-by-case basis if their health status is determined to be stable after consultation with the Medical Monitor.
* Patients with end-stage renal disease receiving hemodialysis via CVC.
* Patients must be expected to receive hemodialysis through a direct or cuffed, tunneled dual lumen catheter or 2 cuffed, tunneled single lumen catheters for a minimum of 45 catheter-days after Day 1.
* Patients must have been receiving dialysis for a minimum of 6 dialysis sessions at the study center dialysis clinic prior to the signing of the Informed Consent Form (ICF).
* Patients must have received dialysis at their prescribed blood flow rate (+/- 10%) for at least 2 consecutive dialysis sessions prior to signing the ICF.
* Patients must have 2 screening pre-pump arterial pressure measurements (collected during the first 20 minutes of dialysis) that differ by less than or equal to (≤) 20 mmHg at 2 consecutive dialysis sessions when receiving dialysis at their prescribed blood flow rate (+/- 10%) prior to randomization.

Exclusion Criteria:

* Clinical signs and/or symptoms of a local or systemic infection within 14 days prior to Day 1.
* Evidence of infection of the catheter exit site/tunnel within 14 days prior to Day 1.
* Patients who have received systemic antibiotics within 14 days prior to Day 1.
* History of fever (T > 37.5°C) or chills within 14 days prior to Day 1.
* An occluded catheter (blood flow inadequate for dialysis) or a catheter that required thrombolytic treatment within 14 days prior to Day 1.
* A catheter coated or impregnated with an antithrombotic, antimicrobial or antiseptic agent, including heparin.
* A catheter coated or impregnated with an antithrombotic, antimicrobial or antiseptic agent, including heparin.
* Catheters that are deemed by their manufacturers to be incompatible with alcohol-containing solutions. These include, but are not limited to:

  1. Angiodynamics - LifeJet® VP VascPak Catheter.
  2. Angiodynamics - Schon™ Chronic Hemodialysis Catheter.
  3. Angiotech - Hemostream™ Chronic Dialysis Catheter.
  4. Bard - all Bard Catheters.
* The use of TEGO® or TEGO-like catheter caps. Patients may be switched to standard catheter caps in order to participate in this study.
* Patients with a known or documented allergy to TMP or TMP-containing drugs, ethanol, ethylene diamine tetraacetic acid (EDTA), propylene glycol and/or glycerin.
* Patients with a history of heparin-induced thrombocytopenia or in whom the use of heparin is contraindicated. (Note: If the use of heparin is restricted for only a specified period of time, the patient may be enrolled at a later date when the use of heparin is no longer contraindicated.)
* Evidence of acute/ongoing hepatic injury (alanine aminotransferase [ALT] > 300 IU/L) or chronic hepatic insufficiency (Total bilirubin > 2.0 mg/dL and/or albumin < 3.0 g/dL during Screening or within 30 days prior to Screening). Note: A patient whose albumin level is low solely due to nephrotic syndrome may be enrolled (with Medical Monitor approval) if the albumin level has been stable for at least 3 months prior to ICF signature.
* Patients who the Investigator believes have a prognosis for survival of less than 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The number of adverse events (AEs), serious adverse events (SAEs) and device deficiencies (DDs) in the experimental and control populations | 39 weeks
The number of thrombolytic treatment events in the experimental and control populations. | 39 weeks
  Thrombolytic treatments may be required to maintain catheter blood flow rates when blood flow is measured under standardized conditions and compared to blood flow at study entry. The number of treatment events in the experimental and control populations is inversely related to the ability of the lock solution to maintain catheter patency.
The number of Central Line Associated Blood Stream Infections (CLABSI events) in the experimental and control populations. | 39 weeks
  CLABSI is defined by the CDC as a documented blood stream infection (bacterial or fungal) in a patient with a CVC with no other source of infection identified by a qualified physician.

SECONDARY OUTCOMES:
The number of Lock Solution Failures in the experimental and control populations. | 39 weeks
  "Lock Solution Failure" is defined as the sum of CLABSI events plus Occlusive Malfunction events. Occlusive malfunction is defined as the inability to return catheter blood flow rates to greater than 80% of baseline blood flow measrued at study entry under standardized conditions after treatment with tissue plasminogen activator (thrombolytic treatment).
The number of Occlusive Malfunction events in the experimental and control populations. | 39 weeks
The number of lock solution aspirate cultures that are positive for bacterial or fungal growth in the experimental and control populations. | 39 weeks
The number of catheters removed from the experimental and control patients that are found to have bacterial or fungal biofilm present inside the catheter lumen(s). | 39 weeks
Catheter blood flow rates measured under standardized conditions over the duration of the study in the experimental and control populations. | 39 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John C Cheronis, MD PhD, Study Director — Great Lakes Pharmaceuticals Inc.
Locations (21):
- Hungary (10):
  - FMC Dialízis Központ Péterfy S. Kórház, Budapest
  - FMC Dialízis Központ Szent István Kórház, Budapest
  - FMC Szépvölgyi Dialízis Központ, Budapest
  - DE OEC Nephrologiai Tanszék, Debrecen
  - FMC Dialízis Központ Eger, Eger
  - FMC Dialízis Központ Kecskemét, Kecskémet
  - FMC Nefrológiai Központ Miskolc, Miskolc
  - FMC Dialízis Központ Pécs, Pécs
  - FMC Szatellita Dialízis Központ Pécs, Pécs
  - Szegedi Tudományegyetem, Szeged
- Poland (11):
  - Stacja Dializ w NZOZ Centrum Chorób Wewnętrzynych "EL-VITA" w Elblągu, Elblag
  - Niepubliczny Zakład Opieki Zdrowotnej Diaverum Gdańsk Kartuska, Stacja Dializ, Gdansk
  - Stacja Dializ NZOZ Diaverum, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Klinika Nefrologii, Transplantologii i Chorób Wewn, Gdansk
  - Stacja Dializ NZOZ Avitum w Legnicy, Legnica
  - Uniw. Szpital Kliniczny im. N.Barlickiego,Oddział Nefrologii, Pododdział Dializ, Lodz
  - Stacja Dializ NZOZ Avitum w Miechowie, Miechów
  - Szpital Kliniczny im. H. Święcickiego, Oddział Nefrologii, Pododdział Dializ, Poznan
  - Radomski Szpital Specjalistyczny im. T. Chałubińskiego, Oddział Dializ, Radom
  - Stacja Dializ NZOZ Diaverum w Tczewie, Tczew
  - Stacja Dializ NZOZ Avitum w Zgierzu, Zgierz

REFERENCES:
- [Derived] Rijnders B, DiSciullo GJ, Csiky B, Rutkowski B, Appelt K, Cheronis J, Aitchison R, Gordon G, Jadoul M, Fluck R. Locking Hemodialysis Catheters With Trimethoprim-Ethanol-Ca-EDTA to Prevent Bloodstream Infections: A Randomized, Evaluator-blinded Clinical Trial. Clin Infect Dis. 2019 Jun 18;69(1):130-136. doi: 10.1093/cid/ciy840. PMID 30281074